CLINICAL TRIAL: NCT05866809
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, 12 Weeks, Therapeutic Exploratory Phase 2 Clinical Study to Evaluate the Safety and Efficacy of HK-660S in Patients With Primary Sclerosing Cholangitis (PSC)
Brief Title: Evaluation of the Safety and Efficacy of HK-660S in Patients With Primary Sclerosing Cholangitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CuromeBiosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HK-660S-201
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-05

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HK-660S (Experimental): Oral administration of HK-660S 100 mg (1 tablet) twice daily before morning and evening meals
  Interventions: Drug: HK-660S
- Placebo (Placebo Comparator): Oral administration of placebo 1 tablet twice daily before morning and evening meals
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HK-660S — Administered orally
  Arms: HK-660S
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the improvement of bile duct strictures following the administration of HK-660S in patients with Primary Sclerosing Cholangitis(PSC). Percentage of subjects who show improvement of severity of PSC as assessed by Magnetic Resonance Cholangiopancreatography(MRCP) at Week 12 from baseline, with improvement defined as a decrease of -1 or more in the MRCP and change of alkaline phosphatase(ALP) level will be assessed at Week 12 from baseline.

DETAILED DESCRIPTION:
Sclerosing cholangitis is a rare, chronic, cholestatic liver disease caused by inflammation and fibrosis of the intrahepatic/extrahepatic biliary tract. Its pathophysiology involves destruction and stricture of the bile duct due to diffuse inflammation and fibrosis of the bile duct. The selected subjects will be randomly assigned to either active or placebo groups and administered 100 mg of HK-660S or placebo (1 tablet) twice a day for 12 weeks. After Visit 2, subjects will visit the study center at Week 4 (Visit 3), Week 8 (Visit 4), Week 12 (Visit 5 / End of Treatment), and Week 16 (Visit 6 / Follow-up) to assess efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 17 years
* Subjects who have a diagnosis of PSC
* Subjects who are able to understand the information provided directly or via his/her representative and give voluntary, written consent to participate in the study.

Exclusion Criteria:

* Subjects with an average alcohol intake of more than 20g per day within 2 years prior to screening.
* Subjects who have a diagnosis of type 1 diabetes or uncontrolled type 2 diabetes (HbA1c ≥ 9%) prior to screening.
* Subjects who have chronic liver diseases other than PSC
* Subjects who have a diagnosis of primary biliary cirrhosis or secondary sclerosing cholangitis in MRCP or Endoscopic Retrograde Cholangiopancreatography(ERCP) prior to screening.
* Subjects who have obstacles to MRCP implementation
* Subjects who have a positive result of hepatitis B surface antigen (HBsAg test) and/or hepatitis C antibody (HCV-Ab test)
* Subjects who have Alanine Aminotransferase(ALT) or Aspartate aminotransferase(AST) > 10 x upper limit of normal(ULN)
* Subjects who have serum creatinine ≥ 2 mg/dl
* Subjects who have weight changes of 5 kg or more within 6 months prior to screening
* Subjects who are deemed unsuitable for participation in the study at Screening, at the discretion of the investigator, due to the following: cirrhosis, severe metabolic disease, severe renal failure, severe lung disease, severe neuro/psychiatric disease, muscle disease, etc.
* Subjects who have any clinically significant cardiovascular diseases
* Subjects who have thyroid diseases including hyperthyroidism and hypothyroidism
* Subjects who have a history of immune diseases
* Subjects who had bariatric surgery within 6 months prior to screening
* Subjects who had liver transplant surgery
* Subjects who have a diagnosis of HIV infection
* Subjects who have a history of chronic infections or have severe or life-threatening infections, or symptoms that may be considered related to infections
* Subjects diagnosed with a malignant tumor without complete cure within 5 years prior to screening
* Subjects whose medication history includes any of the following drugs, within a period of 5 times the half-life of the respective drug prior to screening:

  * Therapeutics agents for steatohepatitis: thiazolidinediones, high-dose vitamin E (800 IU/day), pentoxifylline
  * Medications possibly related to PSC: high-dose ursodeoxycholic acid (UDCA; doses smaller than 23 mg/kg/day may be permitted if administered stably without change in dosage from 3 months prior to screening), immunosuppressants, obeticholic acid (OCA), azathioprine, budesonide, docosahexaenoic acid, methotrexate, metronidazole, minocycline, mycophenolate mofetil, nicotine, pentoxifylline, pirfenidone, prednisolone, systemic glucocorticoids, tacrolimus, vancomycin
* Subjects who administered herbal medicine or folk remedies to improve fatty liver disease within 2 weeks prior to screening
* Subjects who have a history of alcohol or drug abuse within 5 years prior to screening
* Subjects who have a hypersensitivity to any excipients of the study drug
* Subjects who participated in another drug trial within 30 days prior to screening
* Subjects who are considered inappropriate to participate in clinical trials at the discretion of the investigator

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
MRCP | Week 12 from baseline
  Percentage of subjects who show improvement of severity of PSC as assessed by MRCP with improvement defined as a decrease of -1 or more in the MRCP score
ALP | Week 12 from baseline
  Change of ALP level

CONTACTS AND LOCATIONS:
Overall Officials: Do-hyun Park, Principal Investigator — Asan Medical Center
Locations (4):
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - ASAN Medical Center, Seoul
  - Samsung Medical Center, Seoul